CLINICAL TRIAL: NCT02735798
Title: A Pilot Study of 64-Cu Labeled Brain PET/MRI for MM-302, a Novel HER2 Targeting Agent, in Advanced HER2+ Cancer With Brain Metastases
Brief Title: 64-Cu Labeled Brain PET/MRI for MM-302 in Advanced HER2+ Cancers With Brain Mets
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study was not started due to the sponsor choosing to not fund the trial.
Sponsor: Pamela Munster (Other)
Responsible Party: Sponsor-Investigator, Pamela Munster, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15952
Record Dates: First submitted 2016-04-01; First posted 2016-04-13 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Brain Metastases; Documented Her2 Overexpression; Advanced Solid Tumor; Neurologically Stable
MeSH Terms: conditions — Brain Neoplasms | interventions — gancotamab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Study - Arm 1 (Experimental): 10 patients will receive standard imaging at baseline, incl. FDG-PET/CT plus MR brain imaging. Patients will subsequently start protocol therapy with MM-302 and trastuzumab given on day 1 of an every 21-day dosing cycle, at recommended phase 2 dose of 30 mg/m2. Patients will receive 64Cu-labeled MM-302 (3-5 mg/m2 doxorubicin) 3 hours after unlabeled dose of MM-302. Integrated MR/PET imaging of brain and whole body will be performed at 2 time points following 64Cu-labeled MM-302 administration: (1) within 3 hours (+/- 1 hour) of labeled drug injection, and (2) 24 hours (+/- 6 hours) post-injection. Patients will continue to receive doses of unlabeled MM-302 plus trastuzumab every 3 weeks until clinical or radiographic disease progression (in brain or systemically) or unacceptable toxicity, whichever occurs soonest. MRI and FDG-PET/CT scans will be performed every 9 weeks to monitor for treatment response and disease progression.
  Interventions: Drug: MM-302; Drug: Trastuzumab

INTERVENTIONS:
Drug: MM-302
  Other Names: MM-302 brain study
Drug: Trastuzumab
  Other Names: Herceptin

SUMMARY:
This is a single arm pilot study of 64Cu-MM-302 and unlabeled MM-302 in combination with trastuzumab in 10 patients with advanced HER2+ cancer with new or progressive brain metastases. Patients will receive standard imaging at baseline, including FDG-PET/CT plus MR brain imaging. Patients will subsequently start protocol therapy with MM-302 and trastuzumab given on day 1 of an every 21-day dosing cycle, at the recommended phase 2 dose of 30 mg/m2. Patients will receive 64Cu-labeled MM-302 (3-5 mg/m2 doxorubicin) three hours after unlabeled dose of MM-302. Integrated MR/PET imaging of the brain and whole body will be performed at two time points following 64Cu-labeled MM-302 administration: (1) within 3 hours (+/- 1 hour) of labeled drug injection, and (2) 24 hours (+/- 6 hours) post-injection. Patients will continue to receive subsequent doses of unlabeled MM-302 plus trastuzumab every 3 weeks until clinical or radiographic disease progression (either in the brain or systemically) or unacceptable toxicity, whichever occurs soonest. MR brain imaging and FDG-PET/CT scans will be performed every 9 weeks to monitor for treatment response and disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced solid tumor malignancy with documented HER2 overexpression or gene amplification on prior archival tumor tissue by CLIA-certified laboratory
* New or progressive brain metastases with at least one metastasis measuring ≥ 1 cm in longest diameter on MR imaging
* Patients may have extra-cranial metastatic disease but this is not required for study entry
* Neurologically stable as defined by ALL of the following:

  * Stable or decreasing dose of steroids and anti-convulsants for at least 14 days prior to study entry
  * No clinically significant mass effect, midline shift, or impending herniation on baseline brain imaging
  * No significant focal neurologic signs and/or symptoms which would necessitate radiation therapy or surgical decompression in the judgment of the treating clinician
  * Prior radiation therapy for treatment of brain metastases completed at least 4 weeks prior to study entry
* Prior radiation therapy for brain metastases allowed but must have been at least 4 weeks prior to study entry and follow up imaging is not consistent with pseudoprogression in the judgment of treating clinician
* Patients must be ambulatory with ECOG performance status of 0 - 1.
* Adequate organ function, including absolute neutrophil count (ANC) ≥1500 cells/uL, hemoglobin ≥9.0 gm/dL, platelets ≥100,000 cells/uL, estimated creatinine clearance ≥50 mL/min (by the Cockcroft Gault equation), bilirubin <1.5x ULN (unless Gilbert's is suspected), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <1.5x ULN (< 3x ULN if known liver metastases).
* Ejection fraction as assessed by MUGA or echocardiogram > 50%
* Prior cumulative doxorubicin exposure < 300 mg/m2 (or epirubicin equivalent)
* Last dose of prior systemic anti-cancer therapy administered at least 5 half-lives or 4 weeks prior to study entry, whichever is shorter
* No contra-indications to MRI (e.g. pacemaker, aneurysm clips, severe claustrophobia)
* Patients will sign a study-specific IRB-approved consent prior to study entry. Patients must be able and willing to consent and undergo study procedures.
* Age ≥18 years old

Exclusion Criteria:

* Prior treatment with MM-302
* Patients with any class of New York Heart Association (NYHA) CHF or heart failure with preserved ejection fraction (HFPEF)
* Patients with a history of known coronary artery disease or a myocardial infarction within the last 12 months
* Patients with persistently uncontrolled hypertension (systolic BP > 160 mm Hg or diastolic BP > 100 mm Hg) despite optimal medical therapy
* Patients with known unstable angina pectoris
* Patients with a known history of serious cardiac arrhythmias requiring treatment (exception: controlled atrial fibrillation, paroxysmal supraventricular tachycardia)
* Patients with a prolonged QTc interval (≥ 450 ms)
* Patients who previously discontinued trastuzumab due to unacceptable cardiac toxicity
* Patients with a history of LVEF decline to below 50% during or after prior trastuzumab/lapatinib or other HER2 directed therapy.
* Current dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy.
* Any serious and/or unstable pre-existing medical, psychiatric, or other medical condition that could interfere with subject's safety, provision of informed consent, or compliance with study procedures
* Presence of leptomeningeal disease in the absence of parenchymal brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
MM-302 drug penetration into the brain | 3 hours
  by Positron emission tomography-magnetic resonance (MR/PET) imaging

SECONDARY OUTCOMES:
Adverse event | 1 year
  In overall cohort NCI CTCAE v.4.0
Overall response rate | 1 year
  By Revised Assessment in Neuro-Oncology (RANO) criteria
Overall response rate | 1 year
  By Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria
Progession-free survival | 1 year
  In the central nervous system (CNS)
Progession-free survival | 1 year
  Systemically
CNS response rate | 1 year
  In overall cohort
Systemic response rate | 1 year
  In overall cohort
Adverse Event | 1 year
  Treatment with radioactive MM-302
Adverse Event | 1 year
  Treatment with MM-302 and trastuzumab

IPD SHARING:
Plan to Share IPD: Undecided